CLINICAL TRIAL: NCT00911534
Title: A Multicenter Randomized Double-Blind Study to Compare the Efficacy, Safety, and Tolerability of Rabeprazole ER 50 mg With Placebo in Subjects With Symptomatic Gastroesophageal Reflux Disease (sGERD)
Brief Title: Comparing the Efficacy, Safety, and Tolerability of Rabeprazole ER 50 mg With Placebo in Subjects With Symptomatic Gastroesophageal Reflux Disease (sGERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-A001-307
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-11

CONDITIONS: Symptomatic Gastroesophageal Reflux Disease (sGERD)
Keywords: Gastroesophageal Reflux Disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rabeprazole sodium
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rabeprazole sodium — One rabeprazole extended release (ER) 50 mg capsule daily; rescue medication will be provided to subjects to take as needed.
  Other Names: rabeprazole sodium extended release
  Arms: 1
Drug: Placebo — One rabeprazole placebo capsule daily; rescue medication will be provided to subjects to take as needed.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy, safety and tolerability of rabeprazole extended release (ER) 50 mg with placebo in subjects with symptomatic gastroesophageal reflux disease (sGERD).

ELIGIBILITY:
KEY INCLUSION CRITERIA:

Male or female, ages 18 through 75 years will be included in the study. Females should be either of nonchildbearing potential or of childbearing potential. Females of childbearing potential must have negative serum and urine pregnancy tests prior to randomization. Female subjects of childbearing potential must agree to use medically acceptable methods of contraception starting at Visit 1 and throughout the entire study period and for 1 month after the last dose of study drug. Women using hormonal contraceptives must also be using an additional approved method of contraception starting at Visit 1 and throughout the entire study period and for 1 month after the last dose of study drug. Pregnant or lactating females are excluded. Subjects must have a history of heartburn, identified as their main complaint, for 6 months or longer.Subjects must have documentation of a minimum of 5 moderate to severe heartburn episodes, 3 of which occur during the daytime and 1 of which occurs during the nighttime, during the last 7 days before randomization. Subjects must be able to read, write, and understand the language of the symptom dairy.

KEY EXCLUSION CRITERIA:

Subjects will be excluded from the study if they are found to have erosive esophagitis during esophagogastroduodenoscopy (EGD) at Screening, current or a history of esophageal motility disorders, current or a history of Barrett's esophagus, current esophageal strictures or esophagitis (known or suspected to be due to etiology other than GERD such as infection or medications), current or a history of Zollinger-Ellison syndrome and acid hypersecretory conditions, or current gastric or duodenal ulcer. Subjects will be excluded if they are found to have current or a history of cancer, with the exception of fully excised skin basal cell carcinoma, inflammatory bowel disease, a history of esophageal, gastric and duodenal surgery, except simple closure of a perforated ulcer. Subjects will be excluded who require daily use of nonsteroidal anti-inflammatory drugs (NSAIDs), oral steroids (>=20 mg/day prednisone or equivalent), or aspirin (>325 mg/day). Female subjects will be excluded who are pregnant, lactating, or have a positive B-human gonadotropin test at Screening/Baseline. Subjects will be excluded who are known to be human immunodeficiency virus (HIV) positive, have participated in another investigational drug study within 30 days prior to screening or are expected to receive an investigational drug during this trial. Subjects who are unwilling to provide informed consent will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, MD, Study Director — Eisai Inc.
Locations (90):
- United States (90):
  - Athens, Alabama
  - Huntsville, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Encinitas, California
  - Irvine, California
  - Lancaster, California
  - Los Angeles, California
  - Merced, California
  - Oceanside, California
  - Orange, California
  - Pasadena, California
  - Sacramento, California
  - San Diego, California
  - Wheat Ridge, Colorado
  - Bridgeport, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Cape Coral, Florida
  - Hialeah, Florida
  - Miami, Florida
  - New Smyrna Beach, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Zephyrhills, Florida
  - Decatur, Georgia
  - Newnam, Georgia
  - Chicago, Illinois
  - Evansville, Indiana
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Hagerstown, Maryland
  - Hollywood, Maryland
  - Chesterfield, Michigan
  - Troy, Michigan
  - Chaska, Minnesota
  - Mexico, Missouri
  - Butte, Montana
  - Haddon Heights, New Jersey
  - Ocean City, New Jersey
  - Vineland, New Jersey
  - Voorhees Township, New Jersey
  - Great Neck, New York
  - Lake Success, New York
  - Pittsford, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Boone, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Greesnboro, North Carolina
  - High Point, North Carolina
  - Jacksonville, North Carolina
  - Kinston, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Rutherford College, North Carolina
  - Cincinnati, Ohio
  - Gallipolis, Ohio
  - Mentor, Ohio
  - Perrysburg, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Simpsonville, South Carolina
  - Franklin, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Joshson City, Tennessee
  - Nashville, Tennessee
  - Corsicana, Texas
  - Houston, Texas
  - Laredo, Texas
  - Odessa, Texas
  - Overland Park, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - West Valley City, Utah
  - Charlottesville, Virginia
  - Christiansburg, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 305 participants who were enrolled into the study, 300 participants received the study treatment.
Groups:
- Placebo: One placebo capsule, orally, each day for 4 weeks, identical in appearance to the RAB (Rabeprazole) ER (Extended Release) 50mg capsule
- RAB ER 50mg: One RAB ER 50mg capsule, orally, each day for 4 weeks
Period: Overall Study
Arm/Group | Placebo | RAB ER 50mg
Started | 147 (Randomized (treated)) | 153 (Randomized (treated))
Completed | 132 | 137
Not Completed | 15 | 16
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 4 | 1
Not completed — Withdrawal of consent | 1 | 4
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RAB ER 50mg | Total
Number analyzed (Participants) | 147 | 153 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.4 (13.32) | 43.8 (12.35) | 44.1 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 105 | 208
  Male | 44 | 48 | 92

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Average Daily Severity Score of Gastroesophageal Reflux Disease (GERD)-Related Symptoms at Week 4
Description: Participants collected GERD-associated symptoms of daytime heartburn, nighttime heartburn and regurgitation in daily symptom diary. Daytime episodes were defined as those that occurred after arising in the morning until retiring in the evening, and nighttime episodes were defined as those that occurred during the night while sleeping or trying to sleep. The severity score was calculated was based on a 5-point Likert scale ranging from 0 (no symptom) to 4 (very severe symptom); higher scores indicated greater disease activity.
Time Frame: Baseline and Week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | RAB ER 50mg
Number analyzed (Participants) | 147 | 153
Scores on a Scale
  Heartburn (Daytime) | -0.82 (0.65) | -1.22 (0.79)
  Heartburn (Nighttime) | -0.74 (0.72) | -1.17 (0.78)
  Regurgitation | -0.49 (0.62) | -0.74 (0.81)

2. Primary Outcome: Mean Percentage of Diary-Recorded Heartburn-Free Days at Week 4
Description: Participants completed a daily symptom diary. A heartburn-free day was defined as participant report of 'No Heartburn' from nighttime and daytime of the diary for the same day.
Time Frame: Week 4
Population: Intent-to-Treat (ITT) Population - all randomized participants who received at least 1 dose of study drug (n=number of participants with evaluable data)
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Placebo | RAB ER 50mg
Number analyzed (Participants) | 147 | 153
Percentage of Days | 21.23 (26.8) | 41.14 (34.49)

3. Other Pre Specified Outcome: Percentage of Participants With Complete Heartburn Relief
Description: Participants completed a daily symptom diary.
Time Frame: Week 2 and Week 4
Population: ITT (n=number of participants with evaluable data)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | RAB ER 50mg
Number analyzed (Participants) | 147 | 153
Percentage of Participants
  Week 2 (n=147, 148) | 3.4 | 15
  Week 4 (n=147, 148) | 7.5 | 22.2

4. Other Pre Specified Outcome: Time to Achieve First 24-Hour Period Without Heartburn
Description: Participants completed a daily symptom diary.
Time Frame: Baseline to Week 4
Population: ITT
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | RAB ER 50mg
Number analyzed (Participants) | 147 | 153
Days | 14.4 (0.84) | 10.6 (0.92)

ADVERSE EVENTS:
Time Frame: For each participant, from the time participant signed the study consent form until resolution or for up to 30 days after study drug discontinuation, whichever came first.
Description: The analysis was performed using the Safety Analysis Set (SAS) defined as all subjects who received at least 1 dose of study drug and had a postbaseline safety assessment.
Arm/Group | Placebo | RAB ER 50mg
Serious Adverse Events (participants affected / at risk) | 1/147 | 0/152
Other Adverse Events (participants affected / at risk) | 0/147 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | RAB ER 50mg (N=152)
Cholecystitis, acute (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No